CLINICAL TRIAL: NCT03157739
Title: MigraineManager: An Individualized Self-Management Tool for Adolescents With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN001 MigraineManager
Record Dates: First submitted 2017-04-04; First posted 2017-05-17 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Migraine Disorders
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of Optimized Prototype (Experimental): Patients and parents will use MigraineManager to complete assessment measures at baseline and post-treatment (i.e., 2 months after baseline). Answers to these measures will determine what interventions each participant will receive. Data obtained in this phase will be used to make final modifications to MigraineManager for large scale testing.
  Interventions: Behavioral: MigraineManager: Individualized Self-Management Tool

INTERVENTIONS:
Behavioral: MigraineManager: Individualized Self-Management Tool — Answers provided during the online assessment will result in certain intervention recommendations. Once assessments are completed, a treatment plan will be automatically generated for patient and parent guidance.

SUMMARY:
The purpose of the study is to develop, evaluate, and optimize "MigraineManager", the first web-based comprehensive self-management tool for adolescents with migraine, their parents, and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with migraines using current International Classification of Headache Disorders criteria (ICHD-3 beta) for migraine with or without aura
* Patient has headache frequency of 8+ per month
* Access to the internet whether public (e.g., library) or private (e.g., home, personal)
* English fluency for patient, caregiver, and clinician

Exclusion Criteria:

* Diagnosis of pervasive developmental disorder in patient or caregiver as determined by medical chart review
* Diagnosis of serious mental illness (e.g., schizophrenia) in patient or caregiver as determined by medical chart review

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Headache frequency | 15 months
  change in number of days with headache

CONTACTS AND LOCATIONS:
Locations (1):
- Kevin Hommel, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No